CLINICAL TRIAL: NCT02745379
Title: Effect of Buccal Fat Pad Derived Mesenchymal Stem Cells Loaded on Allograft and Platelet-rich Plasma in Maxillary Sinus Augmentation
Brief Title: Effect of Buccal Fat Pad Derived Stem Cells in Maxillary Sinus Augmentation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arash Khojasteh, Associate professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sbmu9212
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Prolactin-Releasing Hormone

ARMS (2):
- BFPSC+ (Experimental): The group receives a combination (DFDBA)+buccal fat pad derived stem cells BFPSC and PRF for sinus augmentation
  Interventions: Procedure: BFPSCs+ DFDBA+ PRF
- BFPSC- (Active Comparator): The group receives a combination of demineralized freeze-dried bone allografts DFDBA (lacking any cells) and PRF for sinus augmentation
  Interventions: Procedure: DFDBA + PRF

INTERVENTIONS:
Procedure: BFPSCs+ DFDBA+ PRF
  Arms: BFPSC+
Procedure: DFDBA + PRF
  Arms: BFPSC-

SUMMARY:
In this study the buccal fat pad derived stem cells (BFPSCs) will be harvested from buccal fat pad tissue of patients receiving maxillary sinus augmentation. In the test group the patients receive a combination of platelet rich fibrin (PRF) and freeze dried bone allograft (FDBA) (SureOss, Hansbiomed, Korea) loaded with BFPSCs. The results will be evaluated by cone beam computed tomography (CBCT)and hematoxylin and eosin staining in 6 months.

DETAILED DESCRIPTION:
The buccal fat pad derived stem cells (BFPSCs) is harvested from buccal fat pad tissues. The BFPSCs will be loaded on freeze dried bone allograft (FDBA) (SureOss, Hansbiomed, Korea). Furthermore, twenty milliliters of the venous blood is obtained, placed and collected in a sterile tube, and centrifuged (GAC medical) for 14 minutes at 2800 rpm (approximately 400 g). Following centrifugation, three layers are separated in the tube: cellular plasma at the top, platelet rich fibrin (PRF) clot in the middle and red blood cells at the bottom of the tube. The PRF clot is separated by a sterile pincette.

The patients in the test group receives BFPSCs loaded on DFDBA with PRF for sinus augmentation and the control group receives combination of PRF and DFDBA (lacking any cells).The results will be evaluated by cone beam computed tomography (CBCT) in 6 months and microscopic evaluation of the biopsies by hematoxylin and eosine staining.

ELIGIBILITY:
Inclusion Criteria:

1. patients with posterior maxillary edentulism
2. pneumatized sinus
3. less than 5mm bone height between the alveolar crest and sinus membrane

Exclusion Criteria:

1. smoking
2. history of malignancy
3. radiation
4. chemotherapy
5. pregnancy
6. systemic diseases contradicting dental and surgical treatments
7. conditions or drugs affecting bone remodeling or bone metabolism and connective tissue
8. allergy to collagen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
amount of regenerated bone | 6 months
  the amount of regenerated bone will be assessed by Image Pro software in CBCT images
amount of regenerated bone | 6 months
  the percent of regenerated bone will be assessed on bone biopsies obtained during implant insertion by H&E staining by microscope

CONTACTS AND LOCATIONS:
Overall Officials: Arash Khojasteh, DMD, OMFS, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- School of Dentristry at Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province, Iran